CLINICAL TRIAL: NCT00522808
Title: A Clinical Pharmacology Study to Determine the Pharmacokinetic , Safety and Tolerability Profile and Antiviral Activity of Multiple Oral Doses of A-831 in Otherwise Healthy Male Hepatitis C Carriers With Compensated Liver Disease
Brief Title: A Study of the PK, Safety and Antiviral Activity of A-831 in HCV Carriers
Acronym: CP104
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Need for re-formulation
Sponsor: Arrow Therapeutics (Industry)
Collaborators: DDS, Dundee (Unknown); David Mutimer, Birmingham (Unknown); Ed Gane, ACS New Zealand (Unknown)
Responsible Party: Julie Dent, Arrow Therapeutics
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CP104
Record Dates: First submitted 2007-08-29; First posted 2007-08-30 (Estimated); Last update posted 2008-09-29 (Estimated); Status verified 2008-09

CONDITIONS: Chronic Hepatitis C
Keywords: HCV; antiviral; PK; Safety
MeSH Terms: conditions — Hepatitis C, Chronic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: A-831

SUMMARY:
The purposes of this study are:

* to determine the safety and tolerability of multiple doses of A-831 at various doses
* to determine how multiple doses of A-831 are distributed through the bloodstream
* to determine if A-831 reduces the amount of Hepatitis C virus in the blood

ELIGIBILITY:
Inclusion Criteria:

* Volunteers will be males of any race aged 18-60 years with a BMI between 18 and 32 kg/m2 at the time of the screening medical
* Volunteers who have given their written informed consent to participate in the study
* Volunteers who are willing and able to comply with the protocol and study procedures
* Volunteers who have a diagnosis of chronic hepatitis C infection and are in good health (other than history of Hepatitis C infection)

Exclusion Criteria:

* Voulnteers with concurrent medical conditions or taking concurrent medications

Ages: 18 Years to 60 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 36 (Estimated)
Dates: Start 2007-08; Primary Completion 2008-03 (Actual); Study Completion 2008-05 (Actual)

PRIMARY OUTCOMES:
Safety
PK
Tolerability
Antiviral activity

CONTACTS AND LOCATIONS:
Overall Officials: Brian Sanderson, Principal Investigator — DDS; David Mutimer, Principal Investigator — WTCRF Birmingham; Edward Gane, Principal Investigator — ACS New Zealand
Locations (3):
- ACS, Auckland, New Zealand
- United Kingdom (2):
  - Birmingham WTCRF, Birmingham
  - DDS, Dundee